CLINICAL TRIAL: NCT06653062
Title: Evaluation of Circulating Tumor Mitochondrial DNA (ct-mtDNA) As a Biomarker for Minimal Residual Disease (MRD) Assessment and Recurrence Monitoring in Hepatocellular Carcinoma (HCC)
Brief Title: Circulating Tumor Mitochondrial DNA (ct-mtDNA) As a Biomarker for Hepatocellular Carcinoma Recurrence Surveillance
Acronym: CCGLC-015
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ze-yang Ding, MD, Prof., Tongji Hospital
Other Study IDs: TJ-IRB202407116
Record Dates: First submitted 2024-10-08; First posted 2024-10-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: MRD; ct-mtDNA; recurrence; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — DNA, Mitochondrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Plasma Samples: Peripheral blood samples collected in EDTA anticoagulant tubes will be processed to separate plasma and blood cells within 4 to 8 hours, optimally within 4 hours post-collection. Plasma samples are stored at -20°C to preserve the integrity of circulating tumor DNA (ctDNA) and other biomarkers.
  Blood Cell Samples: Blood cells separated from the plasma are also stored at -20°C for potential future analysis, including but not limited to, complete blood count, differential analysis, and other cellular markers.
  Tumor Tissue Samples: Tumor tissue samples collected during surgery and biopsy will be preserved to allow for genetic and molecular analysis. These samples are crucial for identifying tumor-specific mitochondrial mutations. Tissue samples are stored in liquid nitrogen tanks or at -70°C to maintain their molecular integrity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Plasma and Tumor Tissue Mitochondrial DNA (mtDNA) Mutation Analysis — Targeted Analysis of Mitochondrial Mutations: Unlike many interventions that may focus on nuclear DNA or general tumor markers, this intervention specifically analyzes mutations within the mitochondrial genome. This focus on mtDNA is based on evidence suggesting that mtDNA mutations are more frequent and may serve as more sensitive indicators of minimal residual disease (MRD) in cancer patients.
  Liquid Biopsy Approach: The intervention utilizes a liquid biopsy technique, which involves the collection and analysis of peripheral blood samples to detect circulating tumor DNA (ctDNA). This non-invasive method contrasts with traditional tissue biopsy interventions, offering a less intrusive approach to monitor disease progression and recurrence.

SUMMARY:
This is a prospective, observational, single-center study. The purpose of this study is to evaluate the efficacy of circulating tumor mitochondrial DNA (ct-mtDNA) in plasma as a biomarker for minimal residual disease (MRD) assessment and recurrence monitoring in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a leading cause of cancer-related mortality worldwide, with a significant proportion of cases occurring in China. Despite advancements in treatment, the prognosis for HCC remains poor due to late diagnosis and high recurrence rates. Minimal Residual Disease (MRD) refers to the presence of residual cancer cells after treatment, which can lead to tumor recurrence. The primary objective of this study is to evaluate the effectiveness of plasma tumor mitochondrial mutations as a biomarker for MRD assessment and recurrence monitoring in patients with HCC. The study hypothesizes that the presence and dynamics of tumor mitochondrial mutations in plasma are associated with the risk of recurrence and overall survival in HCC patients. This is a prospective, observational, single-center study conducted by the Chinese Cooperative Group of Liver Cancer (CCGLC) under the auspices of the Chinese Chapter of International Hepato-Pancreato Biliary Association. The study will involve the collection and analysis of plasma samples from patients with HCC to detect ct-mtDNA mutations before and after treatment. The primary clinical endpoint is the impact of MRD status on progression-free survival (PFS). Secondary endpoints include the influence of treatment on MRD markers, the correlation between post-treatment residual tumor molecular burden and PFS, and the ability of MRD detection to predict recurrence earlier than traditional tumor markers or imaging methods. This study seeks to contribute to the field of HCC management by providing a more precise and personalized approach to MRD assessment and recurrence monitoring. The findings have the potential to improve long-term treatment outcomes and quality of life for patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma (HCC);
* Diagnosis of HCC is according to the American Association for the Study of Liver Diseases or European Association for the Study of the Liver guidelines of HCC management;
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or mRESIST criteria.;
* Expected survival time of 12 weeks or more;
* Signed informed consent form and ability to comply with the study visits and related procedures as stipulated in the protocol.

Exclusion Criteria:

* Patients with other active tumors or severe complications;
* Insufficient tumor tissue for MRD detection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve patients diagnosed with hepatocellular carcinoma (HCC) . The target population for the CCGLC-015 study consists of individuals who meet the following criteria:
  Age: Participants must be 18 years of age or older. Diagnosis: Individuals must have a confirmed diagnosis of HCC. Prognosis: Patients are expected to have a life expectancy of at least 12 weeks, indicating a reasonable prospect for survival following study enrollment.
  Informed Consent: All participants or their legally authorized representatives must provide written informed consent. This ensures they are fully aware of the study, objectives, procedures, potential risks, and benefits, and are willing to comply with the study protocol.
  Compliance: Participants must be capable of and agree to adhere to the study's visit schedule and any related procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | PFS will be assessed from baseline (initiation treatment date) to the first occurrence of disease progression or death, with follow-up assessments at regular intervals up to 2 years post-treatment.
  The primary outcome measure of this study is to evaluate the effect of minimal residual disease (MRD) status, as identified by the presence of tumor mitochondrial DNA (mtDNA) mutations in plasma, on the progression-free survival of patients after treatment for hepatocellular carcinoma. Progression-free survival is defined as the time from the initiation of treatment to the first occurrence of disease progression or death due to any cause, as determined by imaging studies following RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Circulating tumor mtDNA (MRD Marker) | Blood samples for MRD marker assessment will be collected at baseline (immediately before treatment) and at 3-7 days post-treatment.
  This secondary outcome measure aims to assess changes in MRD markers before treatment and at a specific time point shortly after treatment (3-7 days). The analysis will determine the immediate impact of medical intervention on the levels of circulating tumor mtDNA, providing insights into the effectiveness of treatment in removing or reducing MRD.
Correlation Between Post-treatment MRD and PFS | Residual tumor molecular burden will be assessed at the time of post-treatment blood sample collection (3-7 days post-treatment), with PFS being measured from baseline to the first occurrence of disease progression or death, up to 2 years post-treatment.
  This secondary outcome measure will analyze the relationship between the quantity of residual tumor molecular burden, as detected by MRD testing, and the length of progression-free survival. The goal is to determine if a higher molecular burden of residual disease is associated with shorter PFS.
Early Detection of Recurrence Through MRD Monitoring | MRD monitoring will be conducted at regular intervals post-treatment, with the earliest detection of recurrence being the primary focus within the two-year follow-up period (e.g., every 3 months).
  The study will evaluate the ability of MRD detection, based on plasma tumor mtDNA mutations, to predict disease recurrence earlier than traditional tumor markers or imaging methods. This comparison will involve monitoring ctDNA levels over the two-year post-treatment period and comparing the timing of abnormal rises in ctDNA to the detection of recurrence by other means.
Comparison of MRD Detection with Tumor Markers for Early Recurrence Detection | Tumor marker levels and MRD status will be assessed at 3-month intervals post-treatment for up to two years, with the timing of abnormal rises being the critical comparison point.
  This outcome measure will specifically compare the timing of increases in circulating tumor DNA (ctDNA) levels, as detected by MRD testing, to the rises in serum tumor markers (AFP, PIVKA-II) to determine which method can detect recurrence sooner.
Comparison of MRD Detection with Imaging for Early Recurrence Detection | Imaging for disease progression will be performed at 3-month intervals or as clinically indicated (up to 2 years), with ctDNA levels being monitored in parallel to determine the lead time of MRD detection over imaging.
  The study will evaluate whether increases in ctDNA levels, as detected by MRD testing, precede objective disease progression detected by imaging methods, thus serving as an earlier indicator of recurrent disease.
Association of mtDNA Mutational Profile with Clinicopathological Features | The association will be analyzed at baseline and throughout the study duration (up to 2 years), with specific evaluations at 3-month intervals.
  An exploratory analysis will investigate whether specific mtDNA mutational profiles are associated with certain clinicopathological features of the cancer, such as tumor size, differentiation, or stage.
Impact of Maintenance Therapy on Negative MRD Detection Rate | Assessment of the impact of maintenance therapy on MRD detection rate will be conducted at follow-up visits where MRD testing is performed at 6-month intervals after the initial treatment phase for up to two years.
  The study will explore whether patients receiving maintenance therapy after the initial treatment phase have a higher rate of negative MRD detection, suggesting a potential role of MRD in guiding therapeutic decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Ze-yang Ding, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided